CLINICAL TRIAL: NCT01130272
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Dose Ranging, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-27018966 in the Treatment of Patients With Irritable Bowel Syndrome With Diarrhea
Brief Title: Efficacy, Safety, and Tolerability of JNJ-27018966 (Eluxadoline) in the Treatment of Irritable Bowel Syndrome With Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Furiex Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27018966IBS2001
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome with diarrhea; Irritable bowel syndrome; Diarrhea predominant irritable bowel syndrome; Colonic diseases; Colonic diseases, functional; Digestive system disease; Gastrointestinal disease; Intestinal disease; Colonic pseudo-obstruction; Diarrhea; Signs and Symptoms, Digestive
MeSH Terms: conditions — Irritable Bowel Syndrome; Colonic Diseases; Colonic Diseases, Functional; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Colonic Pseudo-Obstruction; Diarrhea; Signs and Symptoms, Digestive | interventions — eluxadoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Eluxadoline 5 mg (Experimental): Eluxadoline 5 mg tablets, orally, twice daily for up to 12 weeks.
  Interventions: Drug: Eluxadoline
- Eluxadoline 25 mg (Experimental): Eluxadoline 25 mg tablets, orally, twice daily for up to 12 weeks. .
  Interventions: Drug: Eluxadoline
- Eluxadoline 100 mg (Experimental): Eluxadoline 100 mg tablets, orally, twice daily for up to 12 weeks.
  Interventions: Drug: Eluxadoline
- Eluxadoline 200 mg (Experimental): Eluxadoline 200 mg tablets, orally, twice daily for up to 12 weeks.
  Interventions: Drug: Eluxadoline
- Placebo (Placebo Comparator): Eluxadoline placebo matching tablets, orally, twice daily for up to 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eluxadoline — Tablets, orally, twice daily.
  Other Names: JNJ-27018966
  Arms: Eluxadoline 100 mg; Eluxadoline 200 mg; Eluxadoline 25 mg; Eluxadoline 5 mg
Drug: Placebo — Matching placebo oral tablets twice daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy, safety, and tolerability of different doses of JNJ-27018966 (eluxadoline) compared with placebo in the treatment of patients with irritable bowel syndrome with diarrhea (IBS-d).

ELIGIBILITY:
Key Inclusion Criteria:

* Patient has a diagnosis of IBS by Rome III criteria with a subtype of diarrhea
* Female patients must be:
* postmenopausal, defined as amenorrhea for at least 2 years at Prescreening,
* surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
* abstinent, or
* if sexually active, be practicing an effective method of birth control.

Key Exclusion Criteria:

* Patient has a diagnosis of IBS by Rome III criteria with a subtype of constipation, mixed IBS, or unsubtyped IBS
* Patient has a history of inflammatory or immune-mediated gastrointestinal (GI) disorders including inflammatory bowel disease (ie, Crohn's disease, ulcerative colitis) and celiac disease
* Patient has a history of diverticulitis within 6 months prior to Prescreening
* Patient has a history of intestinal obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, bariatric surgery, adhesions, ischemic colitis, impaired intestinal circulation (eg, aortoiliac disease), thrombophlebitis of a major vein, or hypercoagulable states.

Other protocol-specific eligibility criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2010-04-28 (Actual); Primary Completion 2011-07-14 (Actual); Study Completion 2011-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (228):
- United States (228):
  - Furiex Research Site, Anniston, Alabama
  - Furiex Research Site, Birmingham, Alabama
  - Furiex Research Site, Dothan, Alabama
  - Furiex Research Site, Huntsville, Alabama
  - Furiex Research Site, Mobile, Alabama
  - Furiex Research Site, Montgomery, Alabama
  - Furiex Research Site, Pell City, Alabama
  - Furiex Research Site, Chandler, Arizona
  - Furiex Research Site, Glendale, Arizona
  - Furiex Research Site, Mesa, Arizona
  - Furiex Research Site, Phoenix, Arizona
  - Furiex Research Site, Tempe, Arizona
  - Furiex Research Site, Tucson, Arizona
  - Furiex Research Site, Jonesboro, Arkansas
  - Furiex Research Site, Little Rock, Arkansas
  - Furiex Research Site, Searcy, Arkansas
  - Furiex Research Site, Sherwood, Arkansas
  - Furiex Research Site, Aliso Viejo, California
  - Furiex Research Site, Anaheim, California
  - Furiex Research Site, Azusa, California
  - Furiex Research Site, Burbank, California
  - Furiex Research Site, Carlsbad, California
  - Furiex Research Site, Encinitas, California
  - Furiex Research Site, Garden Grove, California
  - Furiex Research Site, Inglewood, California
  - Furiex Research Site, Laguna Hills, California
  - Furiex Research Site, Long Beach, California
  - Furiex Research Site, Los Angeles, California
  - Furiex Research Site, Murrieta, California
  - Furiex Research Site, Oakland, California
  - Furiex Research Site, Orange, California
  - Furiex Research Site, Sacramento, California
  - Furiex Research Site, San Carlos, California
  - Furiex Research Site, San Diego, California
  - Furiex Research Site, Colorado Springs, Colorado
  - Furiex Research Site, Denver, Colorado
  - Furiex Research Site, Lakewood, Colorado
  - Furiex Research Site, Littleton, Colorado
  - Furiex Research Site, Thornton, Colorado
  - Furiex Research Site, Bristol, Connecticut
  - Furiex Research Site, Waterbury, Connecticut
  - Furiex Research Site, Aventura, Florida
  - Furiex Research Site, Boca Raton, Florida
  - Furiex Research Site, Bradenton, Florida
  - Furiex Research Site, Brandon, Florida
  - Furiex Research Site, Chipley, Florida
  - Furiex Research Site, DeLand, Florida
  - Furiex Research Site, Delray Beach, Florida
  - Furiex Research Site, Doral, Florida
  - Furiex Research Site, Fort Lauderdale, Florida
  - Furiex Research Site, Hialeah, Florida
  - Furiex Research Site, Inverness, Florida
  - Furiex Research Site, Jacksonville, Florida
  - Furiex Research Site, Jupiter, Florida
  - Furiex Research Site, Kissimmee, Florida
  - Furiex Research Site, Largo, Florida
  - Furiex Research Site, Lauderdale Lakes, Florida
  - Furiex Research Site, Melbourne, Florida
  - Furiex Research Site, Miami, Florida
  - Furiex Research Site, Naples, Florida
  - Furiex Research Site, New Port Richey, Florida
  - Furiex Research Site, New Smyrna Beach, Florida
  - Furiex Research Site, Orlando, Florida
  - Furiex Research Site, Plantation, Florida
  - Furiex Research Site, Port Orange, Florida
  - Furiex Research Site, South Miami, Florida
  - Furiex Research Site, St. Petersburg, Florida
  - Furiex Research Site, Tampa, Florida
  - Furiex Research Site, Atlanta, Georgia
  - Furiex Research Site, Columbus, Georgia
  - Furiex Research Site, Duluth, Georgia
  - Furiex Research Site, Macon, Georgia
  - Furiex Research Site, Marietta, Georgia
  - Furiex Research Site, Newnan, Georgia
  - Furiex Research Site, Rome, Georgia
  - Furiex Research Site, Sandy Springs, Georgia
  - Furiex Research Site, Savannah, Georgia
  - Furiex Research Site, Boise, Idaho
  - Furiex Research Site, Idaho Falls, Idaho
  - Furiex Research Site, Meridian, Idaho
  - Furiex Research Site, Nampa, Idaho
  - Furiex Research Site, Champaign, Illinois
  - Furiex Research Site, Chicago, Illinois
  - Furiex Research Site, Morton, Illinois
  - Furiex Research Site, Anderson, Indiana
  - Furiex Research Site, Bloomington, Indiana
  - Furiex Research Site, Evansville, Indiana
  - Furiex Research Site, Indianapolis, Indiana
  - Furiex Research Site, Lenexa, Kansas
  - Furiex Research Site, Mission, Kansas
  - Furiex Research Site, Overland Park, Kansas
  - Furiex Research Site, Topeka, Kansas
  - Furiex Research Site, Wichita, Kansas
  - Furiex Research Site, Bowling Green, Kentucky
  - Furiex Research Site, Lexington, Kentucky
  - Furiex Research Site, Louisville, Kentucky
  - Furiex Research Site, Metairie, Louisiana
  - Furiex Research Site, Monroe, Louisiana
  - Furiex Research Site, Opelousas, Louisiana
  - Furiex Research Site, Shreveport, Louisiana
  - Furiex Research Site, Annapolis, Maryland
  - Furiex Research Site, Chevy Chase, Maryland
  - Furiex Research Site, Hollywood, Maryland
  - Furiex Research Site, Laurel, Maryland
  - Furiex Research Site, Lutherville, Maryland
  - Furiex Research Site, Prince Frederick, Maryland
  - Furiex Research Site, Rockville, Maryland
  - Furiex Research Site, Boston, Massachusetts
  - Furiex Research Site, Brockton, Massachusetts
  - Furiex Research Site, Hyannis, Massachusetts
  - Furiex Research Site, Springfield, Massachusetts
  - Furiex Research Site, Chesterfield, Michigan
  - Furiex Research Site, Interlochen, Michigan
  - Furiex Research Site, Kalamazoo, Michigan
  - Furiex Research Site, Novi, Michigan
  - Furiex Research Site, Troy, Michigan
  - Furiex Research Site, Chaska, Minnesota
  - Furiex Research Site, Jackson, Mississippi
  - Furiex Research Site, Tupelo, Mississippi
  - Furiex Research Site, City of Saint Peters, Missouri
  - Furiex Research Site, Mexico, Missouri
  - Furiex Research Site, St Louis, Missouri
  - Furiex Research Site, Billings, Montana
  - Furiex Research Site, Bozeman, Montana
  - Furiex Research Site, Bellevue, Nebraska
  - Furiex Research Site, Omaha, Nebraska
  - Furiex Research Site, Henderson, Nevada
  - Furiex Research Site, Las Vegas, Nevada
  - Furiex Research Site, Atco, New Jersey
  - Furiex Research Site, Blackwood, New Jersey
  - Furiex Research Site, Elizabeth, New Jersey
  - Furiex Research Site, Marlton, New Jersey
  - Furiex Research Site, Morristown, New Jersey
  - Furiex Research Site, South Bound Brook, New Jersey
  - Furiex Research Site, Vineland, New Jersey
  - Furiex Research Site, Albuquerque, New Mexico
  - Furiex Research Site, Binghamton, New York
  - Furiex Research Site, Brooklyn, New York
  - Furiex Research Site, Great Neck, New York
  - Furiex Research Site, Mineola, New York
  - Furiex Research Site, New York, New York
  - Furiex Research Site, Boone, North Carolina
  - Furiex Research Site, Chapel Hill, North Carolina
  - Furiex Research Site, Charlotte, North Carolina
  - Furiex Research Site, Fayetteville, North Carolina
  - Furiex Research Site, Greensboro, North Carolina
  - Furiex Research Site, Greenville, North Carolina
  - Furiex Research Site, Harrisburg, North Carolina
  - Furiex Research Site, Hickory, North Carolina
  - Furiex Research Site, High Point, North Carolina
  - Furiex Research Site, Jacksonville, North Carolina
  - Furiex Research Site, New Bern, North Carolina
  - Furiex Research Site, Raleigh, North Carolina
  - Furiex Research Site, Wilmington, North Carolina
  - Furiex Research Site, Winston-Salem, North Carolina
  - Furiex Research Site, Fargo, North Dakota
  - Furiex Research Site, Akron, Ohio
  - Furiex Research Site, Beachwood, Ohio
  - Furiex Research Site, Beavercreek, Ohio
  - Furiex Research Site, Cincinnati, Ohio
  - Furiex Research Site, Cleveland, Ohio
  - Furiex Research Site, Columbus, Ohio
  - Furiex Research Site, Dayton, Ohio
  - Furiex Research Site, Franklin, Ohio
  - Furiex Research Site, Mentor, Ohio
  - Furiex Research Site, Miamisburg, Ohio
  - Furiex Research Site, Springfield, Ohio
  - Furiex Research Site, Wadsworth, Ohio
  - Furiex Research Site, Norman, Oklahoma
  - Furiex Research Site, Oklahoma City, Oklahoma
  - Furiex Research Site, Yukon, Oklahoma
  - Furiex Research Site, Dingmans Ferry, Pennsylvania
  - Furiex Research Site, Hermitage, Pennsylvania
  - Furiex Research Site, Jenkintown, Pennsylvania
  - Furiex Research Site, Lancaster, Pennsylvania
  - Furiex Research Site, Lansdale, Pennsylvania
  - Furiex Research Site, Newton, Pennsylvania
  - Furiex Research Site, Sayre, Pennsylvania
  - Furiex Research Site, Uniontown, Pennsylvania
  - Furiex Research Site, Washington, Pennsylvania
  - Furiex Research Site, Cumberland, Rhode Island
  - Furiex Research Site, East Providence, Rhode Island
  - Furiex Research Site, Warwick, Rhode Island
  - Furiex Research Site, Anderson, South Carolina
  - Furiex Research Site, Columbia, South Carolina
  - Furiex Research Site, Greer, South Carolina
  - Furiex Research Site, Mt. Pleasant, South Carolina
  - Furiex Research Site, Rapid City, South Dakota
  - Furiex Research Site, Bristol, Tennessee
  - Furiex Research Site, Chattanooga, Tennessee
  - Furiex Research Site, Germantown, Tennessee
  - Furiex Research Site, Jackson, Tennessee
  - Furiex Research Site, Johnson City, Tennessee
  - Furiex Research Site, Kingsport, Tennessee
  - Furiex Research Site, Nashville, Tennessee
  - Furiex Research Site, Austin, Texas
  - Furiex Research Site, Bedford, Texas
  - Furiex Research Site, Colleyville, Texas
  - Furiex Research Site, El Paso, Texas
  - Furiex Research Site, Fort Worth, Texas
  - Furiex Research Site, Grand Prairie, Texas
  - Furiex Research Site, Grapevine, Texas
  - Furiex Research Site, Houston, Texas
  - Furiex Research Site, Hurst, Texas
  - Furiex Research Site, Irving, Texas
  - Furiex Research Site, Lake Jackson, Texas
  - Furiex Research Site, Marshall, Texas
  - Furiex Research Site, North Richland Hills, Texas
  - Furiex Research Site, Odessa, Texas
  - Furiex Research Site, Plano, Texas
  - Furiex Research Site, San Antonio, Texas
  - Furiex Research Site, Sugar Land, Texas
  - Furiex Research Site, Webster, Texas
  - Furiex Research Site, Logan, Utah
  - Furiex Research Site, Ogden, Utah
  - Furiex Research Site, Salt Lake City, Utah
  - Furiex Research Site, South Jordan, Utah
  - Furiex Research Site, West Jordan, Utah
  - Furiex Research Site, West Valley City, Utah
  - Furiex Research Site, Alexandria, Virginia
  - Furiex Research Site, Chesapeake, Virginia
  - Furiex Research Site, Christiansburg, Virginia
  - Furiex Research Site, Danville, Virginia
  - Furiex Research Site, Fairfax, Virginia
  - Furiex Research Site, Virginia Beach, Virginia
  - Furiex Research Site, Mill Creek, Washington
  - Furiex Research Site, Madison, Wisconsin
  - Furiex Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Fant RV, Henningfield JE, Cash BD, Dove LS, Covington PS. Eluxadoline Demonstrates a Lack of Abuse Potential in Phase 2 and 3 Studies of Patients With Irritable Bowel Syndrome With Diarrhea. Clin Gastroenterol Hepatol. 2017 Jul;15(7):1021-1029.e6. doi: 10.1016/j.cgh.2017.01.026. Epub 2017 Feb 3. PMID 28167156
- [Derived] Andrae DA, Covington PS, Patrick DL. Item-level assessment of the irritable bowel syndrome quality of life questionnaire in patients with diarrheal irritable bowel syndrome. Clin Ther. 2014 May;36(5):663-79. doi: 10.1016/j.clinthera.2014.04.009. Epub 2014 May 9. PMID 24813429
- [Derived] Dove LS, Lembo A, Randall CW, Fogel R, Andrae D, Davenport JM, McIntyre G, Almenoff JS, Covington PS. Eluxadoline benefits patients with irritable bowel syndrome with diarrhea in a phase 2 study. Gastroenterology. 2013 Aug;145(2):329-38.e1. doi: 10.1053/j.gastro.2013.04.006. Epub 2013 Apr 9. PMID 23583433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 patients were randomized more than once, enrolling at a second (or third) site after discontinuation from the first site. Safety data was analyzed according to the highest dose received. Safety Analysis Set: Highest Dose Level in the Participant Flow reflects the reassignment of patients randomized more than once to the highest dose level arm.
Pre-assignment Details: 807 patients were randomized in the trial. 18 of these patients were enrolled at a site terminated by Furiex, reported to the FDA for potential scientific misconduct, and were excluded from all datasets. All Randomized Patients=789 patients.
Groups:
- Eluxadoline 25 mg: Eluxadoline 25 mg tablets, orally, twice daily for up to 12 weeks.
Period: Overall Study
Arm/Group | Eluxadoline 5 mg | Eluxadoline 25 mg | Eluxadoline 100 mg | Eluxadoline 200 mg | Placebo
Started | 107 | 173 | 169 | 171 | 169
Safety Analysis Set: as Randomized (All participants who received study drug as per randomized dose assignment.) | 105 | 171 | 166 | 167 | 162
Safety Analysis Set: Highest Dose Level (Reflects the reassignment of patients randomized more than once to the highest dose level arm.) | 105 (105 total represents 1 patient in from Placebo arm; 1 patient out to 200 mg arm.) | 170 (170 total represents 2 patients in from Placebo arm; 3 patients out to 200 mg arm.) | 165 (165 total represents 1 patient out to 200 mg arm.) | 172 (172 total represents 1 patient in from 5 mg; 3 patients in from 25 mg;1 patient in from 100 mg arms.) | 159 (159 total represents 2 patients out to 25 mg arm; 1 patient out to 5 mg arm.)
Completed | 48 | 131 | 121 | 103 | 117
Not Completed | 59 | 42 | 48 | 68 | 52
Not completed — Adverse Event | 2 | 5 | 6 | 22 | 7
Not completed — IVRS-confirmed constipation | 0 | 1 | 1 | 2 | 0
Not completed — Rescue medications due to diarrhea | 3 | 5 | 8 | 8 | 6
Not completed — Lack of efficacy- uncontrolled diarrhea | 1 | 1 | 0 | 0 | 2
Not completed — Lack of efficacy-uncontrolled IBS-d pain | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 3 | 5 | 5
Not completed — Lost to Follow-up | 4 | 3 | 4 | 7 | 6
Not completed — Withdrawal by Subject | 4 | 11 | 10 | 9 | 8
Not completed — Physician Decision | 1 | 1 | 0 | 1 | 2
Not completed — Sponsor decision | 6 | 15 | 16 | 13 | 16
Not completed — Study arm discontinued | 38 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eluxadoline 5 mg | Eluxadoline 25 mg | Eluxadoline 100 mg | Eluxadoline 200 mg | Placebo | Total
Number analyzed (Participants) | 107 | 173 | 169 | 171 | 169 | 789
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.00) | 45.5 (11.91) | 43.6 (10.89) | 45.0 (11.65) | 44.5 (12.31) | 44.8 (11.88)
Age, Customized [Number; unit: Participants]
  18 to 25 years | 13 | 11 | 11 | 10 | 11 | 56
  26 to 35 years | 14 | 33 | 31 | 32 | 35 | 145
  36 to 45 years | 21 | 33 | 45 | 37 | 33 | 169
  46 to 55 years | 29 | 54 | 58 | 60 | 52 | 253
  56 to 65 years | 30 | 42 | 24 | 32 | 38 | 166
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 120 | 117 | 119 | 118 | 550
  Male | 31 | 53 | 52 | 52 | 51 | 239
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 90 | 144 | 145 | 147 | 150 | 676
  Black or African American | 12 | 21 | 18 | 18 | 17 | 86
  Asian | 3 | 4 | 3 | 4 | 2 | 16
  American Indian or Alaska Native | 1 | 2 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Other | 1 | 2 | 3 | 2 | 0 | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 13 | 31 | 32 | 22 | 24 | 122
  Not Hispanic or Latino | 94 | 142 | 137 | 149 | 145 | 667
Height [Mean (Standard Deviation); unit: cm] | 167.05 (9.807) | 166.26 (9.523) | 168.38 (9.941) | 167.82 (9.201) | 167.40 (9.725) | 167.40 (9.632)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is the number of participants with available weight data for analysis.
  kg
    number analyzed (Participants) | 107 | 173 | 167 | 166 | 162 | 775
    (all) | 89.10 (23.027) | 83.95 (23.657) | 86.04 (23.796) | 86.53 (21.584) | 86.28 (21.246) | 86.15 (22.671)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Number analyzed is the number of participants with available BMI data for analysis.
  kg/m^2
    number analyzed (Participants) | 107 | 173 | 167 | 166 | 162 | 775
    (all) | 31.88 (7.739) | 30.41 (8.398) | 30.16 (7.059) | 30.71 (7.290) | 30.81 (7.443) | 30.71 (7.595)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Composite Responders Based on Improvements From Baseline in Daily Worst Abdominal Pain and Daily Stool Consistency Scores at Week 4
Description: Composite responders were defined as participants who completed at least 5 out of 7 days with diary entries during the interval of interest and met both of the following criteria: 1) Average daily pain response scores over the past week improved by ≥30% and at least 2 points as compared with the baseline average pain score (average of daily worst abdominal pain the week prior to randomization), 2) Bristol Stool Scale (BSS) score of 3 or 4 on 66% of reported days in the past week. Abdominal pain was assessed on an 11-point scale where: 0=no pain to 10=worst pain imaginable. Stool consistency was assessed using the BSS 7-point scale where: 1=separate hard lumps, 2=sausage shaped but lumpy, 3=sausage-like with cracks on the surface, 4=sausage-like but smooth and soft, 5=soft blobs with clear cut edges, 6=fluffy pieces with ragged edges, and 7=watery with no solid pieces.
Time Frame: Baseline (Week prior to Randomization) to Week 4
Population: Intent to treat (ITT) set was defined as the 754 participants that received at least 1 dose of study drug and had baseline and at least 1 postrandomization daily pain rating and 1 postrandomization Bristol Stool Scale (BSS) rating.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 5 mg | Eluxadoline 25 mg | Eluxadoline 100 mg | Eluxadoline 200 mg | Placebo
Number analyzed (Participants) | 105 | 167 | 163 | 160 | 159
percentage of participants | 12.4 | 12.0 | 11.0 | 13.8 | 5.7
Statistical Analysis 1: Comparison: Eluxadoline 5 mg; Test type: Superiority or Other; p = 0.052, ANCOVA; Odds Ratio (OR) = 2.457, 95% CI 2-sided [0.994 to 6.077]
Statistical Analysis 2: Comparison: Eluxadoline 25 mg; Test type: Superiority or Other; p = 0.041, ANCOVA; Odds Ratio (OR) = 2.383, 95% CI 2-sided [1.036 to 5.478]
Statistical Analysis 3: Comparison: Eluxadoline 100 mg; Test type: Superiority or Other; p = 0.090, ANCOVA; Odds Ratio (OR) = 2.079, 95% CI 2-sided [0.893 to 4.842]
Statistical Analysis 4: Comparison: Eluxadoline 200 mg; Test type: Superiority or Other; p = 0.015, ANCOVA; Odds Ratio (OR) = 2.797, 95% CI 2-sided [1.227 to 6.376]

2. Primary Outcome: Percentage of Participants Who Were Composite Responders Based on Improvements From Baseline in Daily Worst Abdominal Pain and Daily Stool Consistency Scores at Week 12
Description: Composite responders were defined as participants who completed at least 5 out of 7 days with diary entries during the interval of interest and met both of the following criteria: 1) Average daily pain response scores over the past week improved by ≥30% and at least 2 points as compared with the baseline average pain score (average of daily worst abdominal pain the week prior to randomization), 2) Bristol Stool Scale (BSS) score of 3 or 4 on 66% of reported days in the past week. The participant recorded their abdominal pain in a daily diary using an 11-point scale where: 0=no pain to 10=worst pain imaginable. The participant recorded stool consistency in a daily diary using the BSS 7-point scale where: 1=separate hard lumps, 2=sausage shaped but lumpy, 3=sausage-like with cracks on the surface, 4=sausage-like but smooth and soft, 5=soft blobs with clear cut edges, 6=fluffy pieces with ragged edges, and 7=watery with no solid pieces.
Time Frame: Baseline (Week prior to Randomization) to Week 12
Population: ITT analysis set was defined as the 754 participants that received at least 1 dose of study drug and had baseline and at least 1 postrandomization daily pain rating and 1 postrandomization Bristol Stool Scale (BSS) rating.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 5 mg | Eluxadoline 25 mg | Eluxadoline 100 mg | Eluxadoline 200 mg | Placebo
Number analyzed (Participants) | 105 | 167 | 163 | 160 | 159
percentage of participants | 8.6 | 13.2 | 20.2 | 15.0 | 11.3
Statistical Analysis 1: Comparison: Eluxadoline 5 mg; Test type: Superiority or Other; p = 0.449, ANCOVA; Odds Ratio (OR) = 0.719, 95% CI 2-sided [0.306 to 1.689]
Statistical Analysis 2: Comparison: Eluxadoline 25 mg; Test type: Superiority or Other; p = 0.583, ANCOVA; Odds Ratio (OR) = 1.208, 95% CI 2-sided [0.615 to 2.373]
Statistical Analysis 3: Comparison: Eluxadoline 100 mg; Test type: Superiority or Other; p = 0.030, ANCOVA; Odds Ratio (OR) = 2.014, 95% CI 2-sided [1.069 to 3.795]
Statistical Analysis 4: Comparison: Eluxadoline 200 mg; Test type: Superiority or Other; p = 0.326, ANCOVA; Odds Ratio (OR) = 1.395, 95% CI 2-sided [0.717 to 2.716]

3. Secondary Outcome: Change From Baseline in the Weekly Pain Scores
Description: The participant recorded their worst daily pain score in a diary using an 11-point scale where: 0=no pain to 10=worst pain imaginable. The daily scores over the previous week were averaged. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Week Prior to Randomization) to Weeks 4, 8, and 12
Population: ITT analysis set was defined as the 754 participants that received at least 1 dose of study drug and had baseline and at least 1 postrandomization daily pain rating and 1 postrandomization Bristol Stool Scale (BSS) rating. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Eluxadoline 5 mg | Eluxadoline 25 mg | Eluxadoline 100 mg | Eluxadoline 200 mg | Placebo
Number analyzed (Participants) | 105 | 167 | 163 | 160 | 159
scores on a scale
  Baseline | 5.75 (1.541) | 5.91 (1.699) | 6.11 (1.723) | 5.78 (1.477) | 5.87 (1.671)
  Change from Baseline to Week 4: number analyzed (Participants) | 97 | 155 | 143 | 140 | 146
  Change from Baseline to Week 4 | -1.76 (1.964) | -2.11 (1.922) | -2.33 (1.945) | -2.20 (1.874) | -2.09 (2.085)
  Change from Baseline to Week 8: number analyzed (Participants) | 82 | 141 | 132 | 120 | 135
  Change from Baseline to Week 8 | -2.35 (2.105) | -2.54 (2.200) | -2.81 (1.973) | -2.58 (2.099) | -2.54 (2.330)
  Change from Baseline to Week 12: number analyzed (Participants) | 58 | 131 | 124 | 107 | 118
  Change from Baseline to Week 12 | -2.50 (1.979) | -2.57 (2.220) | -3.25 (2.115) | -2.96 (2.138) | -2.65 (2.339)

4. Secondary Outcome: Change From Baseline in Weekly BSS Scores
Description: The patient recorded stool consistency in a daily diary using the BSS 7-point scale where: 1=hard stool to 7=watery diarrhea. The daily scores over the previous week were averaged. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Week prior to Randomization) to Weeks 4, 8, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Eluxadoline 5 mg | Eluxadoline 25 mg | Eluxadoline 100 mg | Eluxadoline 200 mg | Placebo
Number analyzed (Participants) | 105 | 167 | 163 | 160 | 159
scores on a scale
  Baseline | 6.19 (0.445) | 6.24 (0.404) | 6.22 (0.429) | 6.23 (0.420) | 6.20 (0.439)
  Change from Baseline to Week 4: number analyzed (Participants) | 97 | 154 | 143 | 140 | 146
  Change from Baseline to Week 4 | -1.09 (1.095) | -1.17 (1.116) | -1.48 (1.326) | -1.66 (1.266) | -0.99 (1.179)
  Change from Baseline to Week 8: number analyzed (Participants) | 82 | 141 | 132 | 120 | 135
  Change from Baseline to Week 8 | -1.19 (1.125) | -1.39 (1.193) | -1.64 (1.331) | -1.71 (1.373) | -1.19 (1.185)
  Change from Baseline to Week 12: number analyzed (Participants) | 58 | 131 | 123 | 107 | 118
  Change from Baseline to Week 12 | -1.37 (1.206) | -1.41 (1.225) | -1.68 (1.296) | -1.89 (1.317) | -1.27 (1.281)

5. Secondary Outcome: Change From Baseline in the Number of Daily Bowel Movements
Description: Participants recorded the number of bowel movements in a daily diary at the same time each day. The number of daily bowel movements over the previous week were averaged. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Week prior to Randomization) to Weeks 4, 8, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: bowel movements per day
Arm/Group | Eluxadoline 5 mg | Eluxadoline 25 mg | Eluxadoline 100 mg | Eluxadoline 200 mg | Placebo
Number analyzed (Participants) | 105 | 167 | 163 | 160 | 159
bowel movements per day
  Baseline | 4.55 (2.474) | 4.43 (3.155) | 5.13 (3.590) | 4.99 (3.206) | 4.91 (3.567)
  Change from Baseline to Week 4: number analyzed (Participants) | 97 | 155 | 143 | 140 | 146
  Change from Baseline to Week 4 | -1.14 (1.702) | -1.19 (1.673) | -1.71 (1.989) | -2.03 (2.519) | -1.39 (3.096)
  Change from Baseline to Week 8: number analyzed (Participants) | 82 | 141 | 132 | 120 | 135
  Change from Baseline to Week 8 | -1.40 (2.093) | -1.31 (1.607) | -1.85 (1.944) | -2.20 (2.927) | -1.65 (3.423)
  Change from Baseline to Week 12: number analyzed (Participants) | 58 | 131 | 124 | 107 | 118
  Change from Baseline to Week 12 | -1.59 (2.413) | -1.38 (1.727) | -2.13 (2.139) | -2.29 (2.857) | -1.71 (3.599)

6. Secondary Outcome: Percentage of Participants With Response Based on Participants Achieving Prespecified Improvement in Symptoms for at Least 50% of the Time
Description: Responders were participants that met both of the following criteria on the same week for at least 50% of time on study: 1) average of daily pain scores over the past week improved by ≥30% compared with baseline average in pain score, 2) ≥50% reduction in the number of days over the past week with a BSS score ≥5 compared with Baseline. Participants must also have had at least 5/7 days diary entry to be considered a responder for that week. Abdominal pain was assessed on an 11-point scale where a score of 0=no pain to 10=worst pain imaginable. Stool consistency was assessed using the BSS 7-point scale where: 1=separate hard lumps to 7=watery with no solid pieces. Response rates (percentage of participants) are based on model estimates from the logistic regression.
Time Frame: Baseline (Week Prior to Randomization) to Weeks 1-12
Population: ITT Analysis Set; Subjects were included in the interval of Weeks 1-4, Weeks 5-8, or Weeks 9-12 if they received at least 1 dose of study medication within that interval.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 5 mg | Eluxadoline 25 mg | Eluxadoline 100 mg | Eluxadoline 200 mg | Placebo
Number analyzed (Participants) | 105 | 167 | 163 | 160 | 159
percentage of participants
  Weeks 1-12 | 16.5 | 20.2 | 29.7 | 30.6 | 19.0
  Weeks 1-4 | 18.0 | 21.0 | 24.9 | 32.7 | 20.0
  Weeks 5-8: number analyzed (Participants) | 90 | 146 | 137 | 125 | 139
  Weeks 5-8 | 29.3 | 34.4 | 43.0 | 39.3 | 30.3
  Weeks 9-12: number analyzed (Participants) | 72 | 137 | 129 | 109 | 126
  Weeks 9-12 | 29.7 | 34.4 | 49.1 | 50.7 | 31.0

ADVERSE EVENTS:
Time Frame: First dose of study drug and up to and including 7 days after date of the last dose of study drug (Up to 114 days)
Description: Safety population: all patients enrolled who received at least 1 dose of study drug. Nine patients were identified as having been randomized more than once in the study, enrolling at a second (or third) site after discontinuation from the first site. All available data for each patient was included in the Safety Analysis Set and was analyzed according to the highest dose level of treatment received.
Arm/Group | Placebo | Eluxadoline 5 mg | Eluxadoline 25 mg | Eluxadoline 100 mg | Eluxadoline 200 mg
Serious Adverse Events (participants affected / at risk) | 1/159 | 1/105 | 3/170 | 1/165 | 3/172
Other Adverse Events (participants affected / at risk) | 25/159 | 20/105 | 34/170 | 27/165 | 43/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | Eluxadoline 5 mg (N=105) | Eluxadoline 25 mg (N=170) | Eluxadoline 100 mg (N=165) | Eluxadoline 200 mg (N=172)
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Noncardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Appendicitis perforated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | Eluxadoline 5 mg (N=105) | Eluxadoline 25 mg (N=170) | Eluxadoline 100 mg (N=165) | Eluxadoline 200 mg (N=172)
Nausea (Gastrointestinal disorders) | 7 | 6 | 11 | 9 | 18
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 6 | 4 | 13
Vomiting (Gastrointestinal disorders) | 1 | 1 | 7 | 7 | 12
Constipation (Gastrointestinal disorders) | 4 | 2 | 5 | 10 | 6
Sinusitis (Infections and infestations) | 9 | 5 | 4 | 3 | 1
Dizziness (Nervous system disorders) | 4 | 4 | 4 | 5 | 11
Headache (Nervous system disorders) | 6 | 3 | 12 | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.